CLINICAL TRIAL: NCT01826773
Title: A Phase II Open-Labeled Study to Evaluate CardioPET™ as a PET Imaging Agent for Evaluation of Myocardial Perfusion and Fatty Acid Uptake in Subjects With Coronary Artery Disease
Brief Title: CardioPET as PET Imaging Agent to Assess Myocardial Perfusion and Fatty Acid Uptake in Known or Suspected CAD Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fluoropharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CardioPET™ P-02; 2012-002261-36 (EudraCT Number)
Record Dates: First submitted 2013-04-04; First posted 2013-04-09 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Coronary Artery Disease
Keywords: CardioPET; Coronary Artery Disease; Myocardial Perfusion Imaging; Coronary Angiography; Myocardial Fatty Acid Utilization
MeSH Terms: conditions — Coronary Artery Disease | interventions — 9-fluoro-3,4-methyleneheptadecanoic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Stress only CardioPET™ (Experimental): Group I will consist of 15-20 patients and will have CardioPET™ imaging performed with a repeat identical stress component at ≥ 48 hours and ≤ 10 days after the initial stress MPI study. There should be no intervention or change in symptoms between the tests, and the patient must have an angiography scheduled to be performed within 30 days.
  The analysis of the acquired imaging data will determine if CardioPET™ is suitable for identifying myocardial flow defects that were observed in exercise or pharmacologic stress Tc-99m MPI imaging. The goal for this CardioPET™ imaging group is to measure blood flow at near maximal stress.
  Interventions: Drug: CardioPET™
- Rest only CardioPET™ (Experimental): Group II will consist of 15-20 subjects will have undergone either, stress, Tc-99m MPI study or stress-echocardiography indicating ≥2 segments of ischemia. These patients must have been referred and scheduled for coronary angiography. If initial evaluation was performed with stress echocardiography, subjects will have either exercise or pharmacologic stress MPI.
  CardioPET™ imaging in these subjects must be performed ≥ 48 hours and ≤ 10 days from the initial stress (stress MPI or echocardiography) at rest only. An angiography must be scheduled to be performed within 30 days.
  Interventions: Drug: CardioPET™

INTERVENTIONS:
Drug: CardioPET™ — CardioPET™ will be intravenously injected to each subject as a single radio-labeled dose of up to 8 mCi (296 MBq).
  Other Names: trans-9-18F-Fluoro-3,4-Methyleneheptadecanoic Acid; FCPHA (Fluoro CycloPropyl Hexadecanoic Acid)

SUMMARY:
The study is designed to evaluate how safe and how well an investigational imaging product CardioPET™ performs as compared to standard approved imaging products in assessing the function of heart muscle in coronary artery disease patients.

DETAILED DESCRIPTION:
The open label, phase II, multi center, study objectives are as follows:

* To evaluate the diagnostic performance of CardioPET™ in assessing myocardial perfusion as compared to standard Tc-99m myocardial perfusion agents with coronary angiography as the standard of reference for CAD.
* To evaluate the safety of CardioPET™ in known or suspected CAD subjects.
* A secondary objective is to assess fatty acid uptake at rest and following stress.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide written informed consent prior to any study related procedures;
* Male and female subjects over 30 years of age with known or suspected CAD;
* Subjects have been evaluated as having known or suspected CAD by either exercise or pharmacologic MPI or echocardiography with ≥2 segments of ischemia and have been referred to coronary angiography for known or suspected CAD;
* Subjects must be able to complete all evaluations within 30 days of Tc-99m MPI imaging, and must be without any intervention or change in symptoms between the tests.

Exclusion Criteria:

* Past or present use of medications that target fatty acid uptake or metabolism, e.g. Ranexa® (Ranolazine);
* Acute changes in comparison to most recent ECG;
* Suspected acute coronary syndrome;
* Chronic renal failure (Cr > 2.5);
* Anemia (Hgb < 10 within past 2 weeks);
* NYHA Class III or IV Congestive heart failure;
* Severe heart valve disease;
* Any exposure to any investigational drugs or devices, within 30 days prior to imaging study;
* Any acute or unstable physical or psychological disease judged by the Investigators based on medical history or screening physical examination;

Female subjects only:

* Subject that has a positive pregnancy test or is lactating or the possibility of pregnancy cannot be ruled out prior to dosing.
* Females not of child-bearing potential require confirmatory documentation in their medical records or must have a negative pregnancy test within 4 hours prior to receiving the test drug and agree to use an acceptable form of birth control for at least 30 days following CardioPET™ administration.

Male subjects:

* Reliable contraception method from the first injection with the tracer until 3 months after the last injection with the tracer. The following contraceptive method(s) is (are) allowed during the study: Condom.
* If your partner becomes pregnant during the study, you should immediately report this to the investigator.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint- sensitivity and specificity of CardioPET™ | One year
  The aim of this clinical protocol is to study CardioPET™ as a PET imaging agent for evaluation of myocardial perfusion in subjects with known or suspected CAD with a single injection of CardioPET™.
  The primary efficacy endpoint for this phase II study is the sensitivity and specificity of CardioPET™ compared to Myocardial Perfusion Imaging (MPI) using coronary angiography as the standard of reference for the detection of Coronary Artery Disease (CAD).

SECONDARY OUTCOMES:
Primary safety endpoints comparing baseline (pre-injection) values to post-injection values for laboratory testing, electrocardiograms, serial QT, and QTc measurements, physical examinations, vital signs and adverse event assessments | Baseline (pre-injection) values to Post-injection values
  * Laboratory Testing- hematology, serum chemistry and urine analysis
  * Electrocardiograms, Serial QT and QTc measurements
  * Physical Examinations
  * Vital signs-heart rate and systolic and diastolic blood pressure
  * Adverse Event Assessments o

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Gheysens, Professor, Principal Investigator — Nucleaire Geneesunde Gasthuisberg Leuven Hospital, Leuven, Belgium
Locations (5):
- Belgium (5):
  - Dienst Nucleaire Geneeskunde, OLV Ziekenhuis Aalst, Aalst
  - Departement de Cardiologie, CU Saint-Luc, Brussels
  - Service de Medicine Nucleaire, CHU Erasme, Brussels
  - Nucleaire Geneesunde Gasthuisberg Leuven Hospital, Leuven
  - Service de Medicine Nucleaire, Centre Hospitalier Univerisataire de Liege, Belgium, Liège

IPD SHARING:
Plan to Share IPD: Undecided